CLINICAL TRIAL: NCT02786641
Title: Induction Chemotherapy of Docetaxel, Cisplatin and Xeloda in Nomogram-predicted High Risk Locoregionally Advanced Nasopharyngeal Carcinoma
Brief Title: Induction Chemotherapy of TPX in Nomogram-predicted High Risk Locoregionally Advanced Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Fang-Yun Xie, Prof., Sun Yat-sen University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2016-FXY-012-Dept. of RT
Record Dates: First submitted 2016-05-26; First posted 2016-06-01 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: nasopharyngeal carcinoma; induction chemotherapy; concurrent chemotherapy; docetaxel; cisplatin; xeloda; nomogram
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Docetaxel; SSRP1 protein, human; Capecitabine; cisplatin-guanosine adduct

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Active Comparator): low risk NPC treated with concurrent chemoradiotherapy
  Interventions: Radiation: IMRT; Drug: Cisplatin 2
- Group B (Active Comparator): high risk NPC treated with concurrent chemoradiotherapy
  Interventions: Radiation: IMRT; Drug: Cisplatin 2
- Group C (Experimental): high risk NPC treated with induction chemotherapy plus concurrent chemoradiotherapy
  Interventions: Drug: Docetaxel; Drug: Cisplatin 1; Drug: Xeloda; Radiation: IMRT; Drug: Cisplatin 2

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 65mg/m2 in induction chemotherapy
  Other Names: T
  Arms: Group C
Drug: Cisplatin 1 — Cisplatin 75mg/m2 in induction chemotherapy
  Other Names: P
  Arms: Group C
Drug: Xeloda — Xeloda 2000mg/m2 D1-14 in induction chemotherapy
  Other Names: X
  Arms: Group C
Radiation: IMRT — IMRT for all patients
Drug: Cisplatin 2 — Cisplatin 100mg/m2 in concurrent chemotherapy
  Other Names: DDP

SUMMARY:
The investigators aim to evaluate the efficiency and toxicities of induction chemotherapy of docetaxel, cisplatin and xeloda in nomogram-predicted high risk locoregionally advanced nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
All eligible patients receive intensity-modulated radiotherapy (IMRT) with a total dose of 68 Gy or higher in 33 fractions to the primary tumor. Nomogram-predicted low risk patients (Group A) receive concurrent chemotherapy, while nomogram-predicted high risk patients are randomized to receive concurrent chemotherapy (Group B) or induction chemotherapy followed by concurrent chemotherapy (Group C). Induction chemotherapy consists of docetaxel 65 mg/m², D1, cisplatin 75 mg/m², D1 and Xeloda 2000mg/m², D1-14 every 3 weeks for 3 cycles. Concurrent chemotherapy consists of cisplatin 100 mg/m², D1 every 3 weeks for 3 cycles.The primary endpoint is failure-free survival (FFS). Secondary end points include overall survival (OS), locoregional relapse-free survival (LRFS), distant metastasis-free survival (DMFS) and the incidence of grade 3 or higher acute toxicities. All efficacy analyses are conducted in the intention-to-treat population, and the safety population include only patients who receive their randomly assigned treatment.

ELIGIBILITY:
Inclusion Criteria:

* Newly histologically confirmed non-keratinizing (WHO 1991) nasopharyngeal carcinoma.
* Tumor staged as III-IVb (the 2010 UICC/AJCC staging system).
* Karnofsky scale (KPS) ≥ 70.
* Adequate marrow: leucocyte count ≥ 4×10E9/L, hemoglobin ≥ 110g/L and platelet count ≥ 100×10E9/L.
* Normal liver function test: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) and bilirubin ≤ 1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) ≤ 2.5×ULN.
* Adequate renal function: creatinine clearance ≥ 60 ml/min or creatinine ≤ 1.5×ULN.
* Patients must give written informed consent.

Exclusion Criteria:

* Prior malignancy, except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer.
* Pregnancy or lactation (consider pregnancy test in women of child-bearing age and emphasize effective contraception during the treatment period).
* History of previous radiotherapy (except for non-melanomatous skin cancers outside intended radiotherapy volume).
* Prior radiotherapy, chemotherapy or surgery (except diagnostic) to primary tumor or nodes.
* Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose > 1.5×ULN), and emotional disturbance.
* Deficient in dihydropyrimidine dehydrogenase

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
FFS | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hui EP, Ma BB, Leung SF, King AD, Mo F, Kam MK, Yu BK, Chiu SK, Kwan WH, Ho R, Chan I, Ahuja AT, Zee BC, Chan AT. Randomized phase II trial of concurrent cisplatin-radiotherapy with or without neoadjuvant docetaxel and cisplatin in advanced nasopharyngeal carcinoma. J Clin Oncol. 2009 Jan 10;27(2):242-9. doi: 10.1200/JCO.2008.18.1545. Epub 2008 Dec 8. PMID 19064973
- [Background] Lee AW, Ngan RK, Tung SY, Cheng A, Kwong DL, Lu TX, Chan AT, Chan LL, Yiu H, Ng WT, Wong F, Yuen KT, Yau S, Cheung FY, Chan OS, Choi H, Chappell R. Preliminary results of trial NPC-0501 evaluating the therapeutic gain by changing from concurrent-adjuvant to induction-concurrent chemoradiotherapy, changing from fluorouracil to capecitabine, and changing from conventional to accelerated radiotherapy fractionation in patients with locoregionally advanced nasopharyngeal carcinoma. Cancer. 2015 Apr 15;121(8):1328-38. doi: 10.1002/cncr.29208. Epub 2014 Dec 19. PMID 25529384
- [Background] Tang LQ, Li CF, Li J, Chen WH, Chen QY, Yuan LX, Lai XP, He Y, Xu YX, Hu DP, Wen SH, Peng YT, Zhang L, Guo SS, Liu LT, Guo L, Wu YS, Luo DH, Huang PY, Mo HY, Xiang YQ, Sun R, Chen MY, Hua YJ, Lv X, Wang L, Zhao C, Cao KJ, Qian CN, Guo X, Zeng YX, Mai HQ, Zeng MS. Establishment and Validation of Prognostic Nomograms for Endemic Nasopharyngeal Carcinoma. J Natl Cancer Inst. 2015 Oct 14;108(1):djv291. doi: 10.1093/jnci/djv291. Print 2016 Jan. PMID 26467665